CLINICAL TRIAL: NCT06622239
Title: A Randomized, Double-Blinded Clinical Trial to Evaluate the Effects of Naltrexone in Improving Nonsuicidal Self-injurious Behavior
Brief Title: Trial to Evaluate the Effects of Naltrexone in Nonsuicidal Self-injury
Acronym: NiNsSIB
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Whanin Pharmaceutical Company (Industry)
Responsible Party: Principal Investigator, Yong Min Ahn, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AYM-NiNsSIB
Record Dates: First submitted 2024-09-11; First posted 2024-10-02 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-10

CONDITIONS: Nonsuicidal Self-Injury
MeSH Terms: conditions — Self-Injurious Behavior | interventions — Naltrexone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- experimental group (Experimental): naltrexone 50mg
  Interventions: Drug: Naltrexone
- comparison group (Placebo Comparator): placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Naltrexone — naltrexone 50mg for 6 weeks
  Other Names: Revia
  Arms: experimental group
Drug: Placebo — placebo for 6 weeks
  Arms: comparison group

SUMMARY:
The goal of this clinical trial is to learn if naltrexone works to treat nonsuicidal self-injurious behavior in adolescents and adults.

DETAILED DESCRIPTION:
Recruiting participants with nonsuicidal self-injurious behavior and randomizing them to the experiment group and the control group at a 1:1 ratio, the test group administers the experiment drug naltrexone along with the general treatment, and the control group provides a placebo. Clinical evaluation including the frequency of self-injurious behavior is conducted every two weeks. The investigator and participants will double-blinded. Analyze the relationship between changes in clinical symptoms and socio-demographic characteristics, diagnosis, clinical characteristics, and anticipated to discover predictors of treatment effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Age: 16 years of age or older
* Clinical interviews meet DSM-5's nonsuicidal self-injury diagnostic criteria
* Nonsuicidal self-injurious behavior has been observed more than once in the past two months
* Obsessive Compulsive Drinking Scale general craving item 2 or more points (strong desire)
* Self-injurious behavior continues even with 4 weeks of general psychiatric treatment for underlying disease
* Anyone who can independently read and fill out the questionnaire and speak Korean
* Who understand the written consent and voluntarily agree to participate in the study
* Female participants of childbearing age must be negative on urine pregnancy test at screening

Exclusion Criteria:

* currently in psychotic or manic conditions
* currently experiencing serious suicidal thoughts
* history of substance-related disorders including opioid
* do not agree to use very effective contraception from the time of signing the test subject's consent form to the end of study period (non-fertility women and postmenopausal women excluded from the contraception requirements)
* Severe medical conditions (angina pectoris, myocardial infarction, arrhythmia, any cancer that is not in remission, hypothyroidism, hyperthyroidism, diabetes, hepatitis B, hepatitis C, epilepsy, dementia, HIV infection)
* intellectual disability or organic brain damage
* difficulty reading and writing Korean
* taking opioid antagonists (methadone, buprenorphine, etc.)
* on an opiate painkiller
* currently opiate dependence
* acute opiate withdrawal symptoms
* naloxone-induced test is positive or the urine test is positive for opiates
* have been sensitized to this drug
* acute hepatitis, liver failure, severe liver failure
* renal disease
* hypersensitivity reaction to the main ingredient or other ingredients of this drug
* a pregnant woman, a woman who may be pregnant, or a lactating woman
* Since this drug contains lactose, genetic problems such as galactose intolerance, Lapp lactase deficiency, glucose-galactose malabsorption, etc
* active liver disease

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Frequency of nonsuicidal self-injurous behavior | 6 weeks
  Total number of nonsuicidal self-injurous behavior during study period

SECONDARY OUTCOMES:
Deliberate Self-harm Inventory | 6 weeks
  change of NSSI frequency acquired by Deliberate Self-harm Inventory (the outcome of this scale does not have score)
Clinical Global Impressions | 6 weeks
  change of Clinical Global Impressions scale the minimum and maximum values are 1 to 7, higher scores mean worse outcome
Obsessive Compulsive Drinking Scale | 6 weeks
  change of Obsessive Compulsive Drinking Scale the minimum and mixiumum values are 0 to 40, higher scores mean a worse outcome
Eating Disorder Examination-Questionnaire | 6 weeks
  change of Eating Disorder Examination-Questionnaire the minimum and mixiumum values are 0 to 6, higher scores mean a worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: Yong Min Ahn, M.D, Ph.D, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided
undecided yet